CLINICAL TRIAL: NCT02901860
Title: Impact of Shift Work on Risk of Cardiovascular Disease and Diabetes: A Cross-sectional Study
Brief Title: Shift Work and Risk of Cardio-vascular Disease
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 11-0725
Record Dates: First submitted 2016-07-25; First posted 2016-09-15 (Estimated); Last update posted 2023-06-02 (Actual); Status verified 2023-06

CONDITIONS: Shift-Work Sleep Disorder
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — Sleep; Diet

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — All blood samples, with the exception of blood work which is sent to the hospital clinical labs, will be identified only with the subject study code.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Traditional workers: Individuals who work 'traditional" work hours, i.e., 9a-5p.
  Interventions: Other: Sleep, Dietary and Cardio-metabolic Measurements
- Non-traditional workers: Individuals who have work hours outside the usual daytime period
  Interventions: Other: Sleep, Dietary and Cardio-metabolic Measurements

INTERVENTIONS:
Other: Sleep, Dietary and Cardio-metabolic Measurements — At home session: 2-weeks of wrist actigraphy and sleep diaries; a food diary for the three days preceding the lab session; 24-h period of ambulatory blood pressure on a non-work day for participant. Work schedules over a 4-week period will be collected and participants identified as traditional or non-traditional workers.
  Subjects will begin the stay in the research unit in the evening and will remain for about 16-20 hr. Saliva samples will be taken every 30 min from admission until bedtime. Bedtime with polysomnography will be from 11:00pm to 7:00am. Questionnaires will be administered; height, weight and waist/hip circumference and bioimpedance measurement; standard 3-h oral glucose tolerance test and blood tests (CBC, electrolytes, renal, liver and thyroid function , hemoglobin A1c, SHBG levels). For individuals with diabetes only fasting blood samples will be taken.

SUMMARY:
The purpose of this research is to test the hypothesis that those with non-traditional work schedules (e.g. shift workers) have a higher cardio-metabolic risk than those with traditional work schedules (e.g. day workers), and that both accumulated sleep debt and the degree of circadian disruption predict the elevated cardio-metabolic risk. The findings of this research are expected to increase our understanding of physiologic tolerance to non-traditional work schedules and provide the basis for the development of methods for the early detection of adverse health effects and determine coping strategies for the millions of workers with non-traditional work schedules.

ELIGIBILITY:
Inclusion Criteria:

Age 18 and older Full-time workers- working between 7:00 a.m. and 7:00 p.m. employed full time at a medical center.

Non-traditional full-time workers- working between 7:00 a.m. and 7:00 p.m and between 7:00 p.m. and 7:00 a.m., employed full time at a medical center.

Exclusion criteria include:

Acute illness or recent change in medication. Persons employed for less than 3 months at their current job

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
cardio-metabolic risk | Once
  24-h ambulatory blood pressure monitoring and 3-h oral glucose tolerance test

SECONDARY OUTCOMES:
Obesity | Once
  height, weight, BMI and waist/hip circumference and bioimpedance measurement of body fat